CLINICAL TRIAL: NCT00256815
Title: Combination of Weekly Chest Radiotherapy and Oral Navelbine for the Palliation of Advanced Non Small Cell Lung Cancer: A Phase I Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clinical Oncology Research Associates (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hypo 3
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2005-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Hypofractionated chest radiation; Oral Navelbine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Radiation

INTERVENTIONS:
Drug: chemotherapy
Procedure: Radiation

SUMMARY:
The study is designed for subjects whose cancer is too advanced and therefore cannot be operated with the goal of completely removing the cancer. At this stage of the disease, most subjects cannot be cured from the disease, however, treatment can help subjects to live longer and better by keeping the cancer under control. All treatment offered to is primarily pursuing that goal. Subjects at this stage of their disease traditionally receive radiation therapy or chemotherapy, both treatments in succession or both concurrently. Recently, the administration of both methods of treatment concurrently has been employed and indicate somewhat better results. Specifically, a class of chemotherapy agents called Vinca Alakaloids used in combination with radiation therapy appear promising as determined in small studies. The drug Navelbine is part of this class of drugs. This drug is approved as an infusion through the veins. The pill form is under development and will be used in this form in this treatment program.

For this protocol, radiation will be administered using a schedule which is more convenient for patients, by once weekly chest irradiation for a total of 12 weeks. Use of this schedule was determined to be as good as the more commonly used daily radiotherapy. The once weekly schedule is less cumbersome as it involves less visits. The rationale and reason why you are being asked to participate in this program is to study whether the drug Navelbine can be given together with the once weekly radiation schedule. Radiation will be administered in two fractions, 6 hours apart on one day. For this program, the drug Navelbine would be made available as a pill, and would not have to be infused through the vein. The proposed protocol will use increasing doses of the drug Navelbine in pill form to find the highest dose of Navelbine that is tolerated in conjunction with radiation therapy. Initially, each subject will receive one dose of Navelbine, which is higher than the dose of the previous subject. This escalation will continue until the highest tolerated dose has been determined.

The administration via pill would be easier and avoid previously experienced side effects that were experienced by infusion into the veins of subjects, such as burning and sores at the infusion site.

DETAILED DESCRIPTION:
35 patients with advanced NSCLC will be enrolled (stages III and IV) and treated once per week in two fractions for a total of 12 cycles using a previous prescription developed by Salazar et al to a total of 6000 rad.

Treatment will be given to a large field with a 2-3 cm tumor margin. All involved or suspicious nodal areas will be radiated as well. The drug Navelbine will be given in a dose escalation on the same day the radiation is administered. The starting dose for Navelbine will be 20 mg/m2 and the escalation will be in 10 mg increments.

ELIGIBILITY:
Inclusion Criteria

1. Pathologically or cytologically confirmed NSCLC. Histology may include adenocarcinoma, squamous cell, large cell undifferentiated, but no bronchoalveolar carcinoma, small cell or carcinoid.
2. Locally advanced NSCLC disease (Stage IIIa or IIIb) or metastatic disease (Stage IV)
3. ECOG performance status 0-2 (See Appendix 1 )
4. Age > 18 years.
5. Absoloute neutrophil count > 1500 / mm3 ,platelet count > 100,000/ mm3
6. Serum bilirubin < upper limit of normal (ULN); ALT and AST < 2.5 X ULN if alkaline phosphatase is < ULN. Alkaline phosphatase may be up to 4 X ULN if transaminases are < ULN.
7. Normal serum creatinine (less than 1.5 mg/dl) or creatinine clearance greater than 30 ml/minute (Cockroft and Gault).
8. No history of allergy to the agents being used in this study.
9. If female of childbearing potential, pregnancy test is negative and must be practicing approved methods of birth control. (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of nonchildbearing potential).
10. If fertile, the patient agrees to use acceptable methods to avoid pregnancy for the duration of the study.
11. No evidence of CHF, ischemic heart disease (NYHA Class III or IV), or serious arrhythmias or recent history of myocardial infarction.
12. No evidence of active infection or serious concurrent medical illness which would jeopardize the ability of the patient to receive with reasonable safety the chemotherapy and radiation program outlined in this protocol.
13. Should a second malignancy be present or discovered, subjects will only be eligible if the NSCLCA is determined by the PI to be the more life-threatening disease compared to the other malignancy in regards of life-expectancy.
14. Patients should have at least a predicted FEV1 of 30%.
15. Signed informed consent has been obtained (see the informed consent form Appendix 2). Each patient must be aware of the neoplastic nature of his/her disease and willingly consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.

3.B. Exclusion Criteria Patients meeting any of the following criteria will not be eligible for the study.

1. Patients with medically uncontrollable hypercoaguability syndromes are not eligible. Patients who are on therapeutic anticoagulation are not excluded.
2. Patients with weight loss > 10% in previous 3 months.
3. Patients with prior Vinca Alkaloid treatment.
4. Subjects where studies or clinical examination demonstrates lack of physical integrity of the upper gastrointestinal tract (e.g. previous significant surgical resection), inability to swallow capsules intact, dysphagia, or those who have malabsorption syndrome.
5. Subjects who have had an organ allograft.
6. Patients with known adverse effects to Vinca Alkaloids.
7. Subjects with several renal impairment (creatinine clearance below 30ml/min [Cockroft and Gault]).
8. Pregnant women and nursing mothers.
9. Sexually active males unwilling to practice contraception during the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 2003-03; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Safety
Toxicity

SECONDARY OUTCOMES:
Efficacy
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Paul Schwarzenberger, MD, Principal Investigator — LSUHSC
Locations (1):
- LSUHSC, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Schwarzenberger P, Theodossiou C, Barron S, Diethelm L, Boyle M, Harrison L, Wynn RB, Salazar OM, Fariss A. Dose escalation of docetaxel concomitant with hypofractionated, once weekly chest radiotherapy for non-small-cell lung cancer: a phase I study. Am J Clin Oncol. 2004 Aug;27(4):395-9. doi: 10.1097/01.coc.0000131943.02929.ac. PMID 15289734
- [Background] Iaffaioli RV, Caponigro F, Tortoriello A, Facchini G, Ravo V, Maccauro M, Dimitri P, Crovella F, Muto P. Accelerated split-course (type B) thoracic radiation therapy plus vinorelbine/carboplatin combination chemotherapy in stage III inoperable non-small cell lung cancer. Eur J Cancer. 1996 Oct;32A(11):1901-4. doi: 10.1016/0959-8049(96)00203-1. PMID 8943672
- [Background] Slawson RG, Salazar OM, Poussin-Rosillo H, Amin PP, Strohl R, Sewchand W. Once-a-week vs conventional daily radiation treatment for lung cancer: final report. Int J Radiat Oncol Biol Phys. 1988 Jul;15(1):61-8. doi: 10.1016/0360-3016(88)90347-1. PMID 2839442
- [Background] Salazar OM, Slawson RG, Poussin-Rosillo H, Amin PP, Sewchand W, Strohl RA. A prospective randomized trial comparing once-a-week vs daily radiation therapy for locally-advanced, non-metastatic, lung cancer: a preliminary report. Int J Radiat Oncol Biol Phys. 1986 May;12(5):779-87. doi: 10.1016/0360-3016(86)90036-2. PMID 3519551